CLINICAL TRIAL: NCT02377713
Title: A Phase 1 Randomized, Double-blind, Placebo-controlled, Single Ascending Dose Study of KHK6640 in Japanese Patients With Alzheimer's Disease.
Brief Title: A Single Dose Study of KHK6640 in Japanese Patients With Alzheimer's Disease.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Kyowa Kirin Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 6640-002
Record Dates: First submitted 2015-02-25; First posted 2015-03-04 (Estimated); Last update posted 2016-12-07 (Estimated); Status verified 2016-12

CONDITIONS: Alzheimer's Disease
Keywords: KHK6640; Phase 1; Japanese; single dose; Alzheimer's disease
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- KHK6640 (Experimental): KHK6640
  Interventions: Drug: KHK6640
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: KHK6640 — Single ascending dose administration
  Arms: KHK6640
Drug: Placebo — Single ascending dose administration
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability and pharmacokinetics of KHK6640, given as a single dose in Japanese patients with Mild to Moderate Alzheimer's Disease.

ELIGIBILITY:
Inclusion Criteria:

* Patients with mild to moderate Alzheimer's Disease
* Body weight ≥ 40 kg and < 100 kg
* Clinical Dementia Rating (CDR) score of 1 or 2
* Mini Mental State Examination (MMSE) score of ≥ 17 amd ≤ 26

Exclusion Criteria:

* Previous active treatment with an Alzheimer's Disease immunotherapy in an investigational study
* Use of another investigational drug within 4 months prior to the enrollment
* Subjects who meet National Institute of Neurological Disorders and Stroke/Association Internationale pour la Recherche et l'Enseignement en Neurosciences (NINDS/AIREN) criteria for vascular dementia
* Subjects with a history of presence of clinically significant seizures, brain trauma, transient ischemic attack, and/or cerebrovascular disease
* Subjects with a presence of a neurological condition that could be contributing to cognitive impairment above and beyond that caused by the subject's Alzheimer's Disease
* Subjects who have evidence of infection, tumor, or other clinically significant lesions that could indicate a dementia diagnosis other than Alzheimer's Disease

Ages: 55 Years to 84 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2015-03; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | Up to 90 days

CONTACTS AND LOCATIONS:
Locations (1):
- Tokyo, Sumida-ku, Japan